CLINICAL TRIAL: NCT02184793
Title: Impact of an Electronic Monitoring Device on Maintaining a Correct Elevation of Head of Bed for Mechanically-ventilated Patients in Intensive Care Unit
Acronym: Inclinometre2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: P080407
Record Dates: First submitted 2014-06-25; First posted 2014-07-09 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Mechanically-ventilated Patients
Keywords: mechanical ventilation; semirecumbent position; electronic monitoring device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMD (Inclinomax) then usual care (Other): EMD (electronic monitoring device) : recording the head of bed inclination degree with digital display and alarm on for 24h.
  Usual care : recording the head of bed inclination degree with masked digital display and alarm off for 24h.
  Interventions: Device: EMD (Inclinomax)
- usual care then EMD (Inclinomax) (Other): Usual care : recording the head of bed inclination degree with masked digital display and alarm off for 24h.
  EMD (electronic monitoring device) : recording the head of bed inclination degree with digital display and alarm on for 24h.
  Interventions: Device: EMD (Inclinomax)

INTERVENTIONS:
Device: EMD (Inclinomax) — EMD (electronic monitoring device) : recording the head of bed inclination degree with digital display and alarm on
  Other Names: EMD (electronic monitoring device)

SUMMARY:
Maintaining mechanically-ventilated patients in semi-recumbent position (defined by a head of bed inclination between 30° and 45°) would decrease the risk of pneumopathy occurrence in those patients. However, such a bed inclination frame is still difficult to maintain in day-to-day care.

The aim of the study is to evaluate the impact of an electronic monitoring device on the proportion of time spent per day in semi-recumbent position, as defined by a head of bed inclination between 40° and 50°, in mechanically-ventilated patients.

DETAILED DESCRIPTION:
Maintaining semi-recumbent position (defined by a head of bed inclination between 40° and 50°) is an international guidance to prevent ventilator-associated pneumopathy which is the main nosocomial infection in intensive care unit. However, maintaining such an inclination has been shown to be difficult in day-to-day care.

This could be improved by using an assistance device that would measure inclination of the head of bed in real time and trigger an alarm when the value order is not reached, hence allowing a quick readjustment if necessary.

The investigators want to evaluate en electronic monitoring device (EMD) that is removable and adjustable to all beds, which would allow a whole intensive care unit to be fully equipped at low cost.

Hypothesis : using an EMD could improve the proportion of time spent per day in semi-recumbent position (defined by a head of bed inclination between 40° and 50°) in mechanically-ventilated patients.

Primary objective : to evaluate the impact of an EMD with alarm on the proportion of time spent per day in semi-recumbent position, as defined by a head of bed inclination between 40° and 50°, in mechanically-ventilated patients.

Secondary objectives :

* to evaluate the impact of the EMD on the head of bed inclination overall mean
* to evaluate the impact of the EMD on the proportion of time spent per day with a head of bed inclination superior to 30°
* to evaluate the impact of the EMD on the proportion of time spent per day with a head of bed inclination between 30° and 45°
* to study factors associated to a head of bed inclination inferior to 30° for more than 12hrs per 24hrs

ELIGIBILITY:
Inclusion Criteria:

* patient with invasive mechanical ventilation
* expected mechanical ventilation duration for more than 48h after inclusion
* signature of an informed consent by a relative
* patient affiliated to a social security scheme (beneficiary or assignee)

Exclusion Criteria:

* age<18 years old
* mechanical ventilation with tracheotomy
* contraindication to semirecumbent position (e.g., spinal cord injury, important sacral bedsore, counterpulsation balloon, femoral cannulation for extracorporeal circulation) or expected indication to another position within the following 48 h after inclusion (e.g., ventral decubitus for hypoxemia pulmonary pathology)
* SAPS II score > 65 at the admission (moribund patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
proportion of time spent per day in semirecumbent position as defined by a head of bed inclination between 40° and 50° | 24hrs
  head of bed inclination recording during 24h

SECONDARY OUTCOMES:
head of bed inclination overall mean | 24hrs
  head of bed inclination recording during 24h
proportion of time spent per day with a head of bed inclination superior to 30° | 24hrs
  head of bed inclination recording during 24h
proportion of time spent per day with a head of bed inclination between 30° and 45° | 24hrs
  head of bed inclination recording during 24h

CONTACTS AND LOCATIONS:
Overall Officials: Lila Bouadma, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat Claude Bernard, Paris, France